CLINICAL TRIAL: NCT06164041
Title: Training and Detraining Effects of a Ten-week Physical Activity Program Implemented Through Mobile Applications on Body Composition and Fitness of Adolescents Aged 12-16 Years.
Brief Title: Training and Detraining Effects of a Physical Activity Program Implemented Through Mobile Applications in Adolescents.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Raquel Vaquero-Cristóbal, Principal Investigator, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MobileApps-Re
Record Dates: First submitted 2023-11-22; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Adolescent Behavior; Mobile Applications; Physical Activity; Physical Condition; Body Composition
MeSH Terms: conditions — Adolescent Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control Group (No Intervention): The control group did not use any of the research mobile applications, but were measured at pre, post and post 2. They continued attending physical education classes normally and practicing their sports activities.
- Cardiovascular training through the application "MapMyWalk" (Experimental): The adolescents who used this application were required to record their weekly workouts. To do this, before starting the workout, they entered the application, selected "walking" and started the record. The application included different warnings and alerts to encourage the practice of physical activity. Each week they had to make a weekly report with the distance covered.
  Interventions: Behavioral: The use of mobile applications promoted from the physical education classroom to improve adolescent health.
- Cardiovascular training through the application "Strava" (Experimental): The adolescents who used this application were required to record their weekly workouts. To do this, before starting the workout, they entered the application, selected "walking" and started the record. The application included different warnings and alerts to encourage the practice of physical activity. Each week they had to make a weekly report with the distance covered.
  Interventions: Behavioral: The use of mobile applications promoted from the physical education classroom to improve adolescent health.
- Cardiovascular training through the application "Pacer" (Experimental): The adolescents who used this application were required to record their weekly workouts. To do this, before starting the workout, they entered the application, selected "walking" and started the record. The application included different warnings and alerts to encourage the practice of physical activity. Each week they had to make a weekly report with the distance covered.
  Interventions: Behavioral: The use of mobile applications promoted from the physical education classroom to improve adolescent health.
- Cardiovascular training through the application "Pokémon Go" (Experimental): This application is considered immersive as teenagers enter a virtual world. In it, the distance traveled in the real world was accounted for in the video game, also appearing different Pokémon that they could capture, making the gaming experience more playful. In the same way, the teenagers had to keep a weekly record of the distance traveled.
  Interventions: Behavioral: The use of mobile applications promoted from the physical education classroom to improve adolescent health.

INTERVENTIONS:
Behavioral: The use of mobile applications promoted from the physical education classroom to improve adolescent health. — Before starting the intervention, a total of 465 adolescents participated in pretest measurements (T1).
  Researchers in charge of explaining how the apps worked were not involved in the measurements or subsequent analysis, as they knew which student belonged to each App and control group. Once each app had been described and its use explained, a training plan was drawn up to be followed during the period of mandatory use.
  The adolescents were motivated to utilize the app for a duration of ten weeks, aiming for a minimum usage of three times per week.
  After the mandatory intervention with the mobile apps, post-test measurements were carried out (T2). Then, a period of 10 weeks was provided in which the use of the app was neither mandatory nor promoted from the physical education subject, after which the post-test 2 measurements (T3) were taken.
  Arms: Cardiovascular training through the application "MapMyWalk"; Cardiovascular training through the application "Pacer"; Cardiovascular training through the application "Pokémon Go"; Cardiovascular training through the application "Strava"

SUMMARY:
The use of mobile applications to promote the practice of physical activity has begun to be used in the adolescent population in recent years. This has made it possible to carry out interventions inside and outside the educational setting, the latter being the ones that have brought the greatest benefits. Thus, it has been observed that the promotion of the use of mobile applications in out-of-school hours from the subject of physical education has reported significant benefits on body composition and fitness in the adolescent population. However, there is no known research that has analyzed whether the effect achieved with mobile applications when their use is mandatory disappears when they are no longer promoted from the physical education subject. Therefore, this project goes further and tries to find out whether after the ten-week period of mandatory use of the applications, adolescents continue to use the applications autonomously and the beneficial effects achieved are maintained or disappear due to the lack of use.

For this purpose, a 10-week intervention was planned in which the adolescents used the mobile applications. Prior to the start of the intervention, the adolescents' body composition and fitness (pre) were measured. At the end of the intervention of mandatory use of the mobile applications, the adolescents were measured again (post). And after the post measurement, the adolescents were left for 10 weeks during which they could use the applications autonomously. A third measurement of the adolescents was performed after this 10-week period (post 2).

The aim of this project was to find out the effects of stopping the use of the mobile fitness apps on body composition and fitness of the adolescents.

ELIGIBILITY:
Inclusion Criteria:

* enrollment in one of the selected educational centers.
* age comprised between 12-16 years old.
* completion of all questionnaires and physical tests during the three measurement periods (T1, T2 and T3).
* attending the kinanthropometric and body composition measurement periods.
* absence of any pathology or injury that would hinder participation in the tests or measurements conducted.

Exclusion Criteria:

* missing more than 20% of the compulsory physical education sessions throughout the academic year.
* lack of mobile phone.
* failure to meet the minimum mandatory weekly distance requirement in the App group when app usage was obligatory.
* changing schools or class group during the course of the intervention.
* starting or ending any form of physical activity during the intervention that could alter the level of physical activity practiced for reasons unrelated to the study.
* having presented any illness during the follow-up period that would have prevented them from engaging in their usual physical activity.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 357 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Physical Activity Level (International Physical Activity Questionnaire for Adolescents) | Through study completion, an average of 1 year
  The Physical Activity Questionnaire for Adolescents will be used to establish the level of sports practice of the adolescents. This questionnaire includes eleven questions related to the practice of physical activity in school, after school, household chores and travel. The questionnaire makes it possible to classify adolescents as inactive or active (light, moderate or vigorous intensity).
Physical condition (Maximal oxygen consumption) | Through study completion, an average of 1 year
  The 20-m shuttle run test evaluates maximal aerobic capacity by means of an incremental 20-meter out-and-back test. The initial speed of the test is 8.5 km/h and is increased every minute by an audible signal. The test ends when the subject stops or fails to reach the reference line two consecutive times. The speed recorded is the speed reached in the last stage that the subject is able to complete. Through the equations of Leger et al. the reference value of the subject's VO2 max. is obtained.
Physical condition (Lower extremity muscle strength) | Through study completion, an average of 1 year
  The countermovement jump test (CMJ) will be used to measure this variable. This test provides information on the explosive strength of the lower body. The CMJ is a vertical jump that begins with the subject in a standing position, followed by knee flexion to a position of approximately 90 degrees, and a rapid extension of the knees to perform a jump in which the maximum height is reached. It should be noted that there is no stop in the knee flexion position since the intention is to take advantage of the explosive elastic reflex energy of the movement. The subjects will perform two repetitions of the jump 2 minutes apart. A MuscleLab force platform (Ergotest Innovation S.A., Norway) will be used to record the data, which will measure the time of flight from the time the subject takes off from the platform to the time the subject re-enters contact with the platform.
Physical condition (abdominal strength) | Through study completion, an average of 1 year
  To assess abdominal muscle endurance will be use Curl-up. The highest number of repetitions the subject completes in one minute will be recorded.
Physical condition (upper extremity muscle strength) | Through study completion, an average of 1 year
  To assess upper limb strength will be used Push-up test. The subject will perform as many repetitions as possible in one minute, or until reaching exhaustion.
Anthropometric Variables (Height) | Through study completion, an average of 1 year
  To measure height, a SECA measuring rod should be used. Adolescents should stand barefoot with their backs against the measuring rod, heels of their feet together and their gaze straight ahead. Measurements will be obtained in centimeters and will be repeated 2 times for each subject. A third measurement will only be taken if the difference between the first and second measurement is greater than 1%.
Anthropometric Variables (Weight) | Through study completion, an average of 1 year
  A Tanita BC 418-MA Segmental scale (Tanita, Tokyo) will be used to measure body weight. The subject will step on the scale with both feet inside the scale and looking straight ahead, without leaning the body. Values will be obtained in kilograms and two measurements will be carried out on each subject. If the difference between both measurements is greater than 1%, a third measurement will be taken.
Anthropometric Variables (Fat mass) | Through study completion, an average of 1 year
  To obtain the fat mass, it will be necessary to previously measure the triceps, thigh and calf folds, and the waist, hip, relaxed arm, thigh and calf perimeters. For these previous measurements, two measurements will be taken in each subject, and a third measurement will be necessary if the difference between the first two is greater than 5%. Once the values of the previous measurements have been obtained, the fat mass can be calculated using the formula of Slaughter et al.
Anthropometric Variables (Fat-free mass) | Through study completion, an average of 1 year
  To obtain the fat-free mass, it will be necessary to previously measure the triceps, thigh and leg folds, and the perimeters of the waist, hip, relaxed arm, thigh and leg. For these previous measurements, two measurements will be taken in each subject, and a third measurement will be necessary if the difference between the first two is greater than 5%. Once the values of the previous measurements have been obtained, the-fat free mass can be calculated using the formula of Poortmans et al.
Anthropometric Variables (BMI) | Through study completion, an average of 1 year
  Previously obtained height and weight measurements will be used to establish the BMI. The formula used will be weight/height^2, and the result will be obtained in kg/m^2. This index is commonly used and is related to metabolic and cardiovascular diseases in adolescents and adults.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica de Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mateo-Orcajada A, Vaquero-Cristobal R, Mota J, Abenza-Cano L. Physical Activity, Body Composition, and Fitness Variables in Adolescents After Periods of Mandatory, Promoted or Nonmandatory, Nonpromoted Use of Step Tracker Mobile Apps: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2024 Jul 30;12:e51206. doi: 10.2196/51206. PMID 39079110